CLINICAL TRIAL: NCT01027637
Title: In Situ Elasticity of Alloderm® in Breast Reconstruction
Brief Title: Regenerative Tissue Matrix for Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: AamirSiddiqui, MD, Division of Plastic Surgery, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HFHS-PS1209; PS1209 (Other Grant/Funding Number: Lifecell)
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; tissue expander; Alloderm; tissue matrix
MeSH Terms: conditions — Breast Neoplasms | interventions — Alloderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alloderm reconstruction (Experimental): All patients recieving the intervention Alloderm for breast reconstruction
  Interventions: Other: 5 mm vessel clips

INTERVENTIONS:
Other: 5 mm vessel clips — evenly placed vessel clips placed at surgery and tracked by ultrasound
  Other Names: Alloderm; acellular regenerative tissue matrix

SUMMARY:
The purpose of this study is to evaluate the role of Alloderm tissue regenerative matrix used in many breast reconstruction operations. When this material is used in the abdomen it often stretches and sometimes needs to be replaced. Although we see good clinical results when used for breast reconstruction, there is no research regarding if or how the material changes in this location. The Alloderm is placed in the breast at the time the expander is placed, post-mastectomy. The expansion is started at the time of surgery and completed during a series of office visit. This process stretches the skin, underlying muscle and presumably the Alloderm. The goal of this study is to better understand the natural history of this material when used for breast reconstruction.

Our objective is to measure changes in the dimension of the tissue matrix material after it has been placed in the breast. These objective findings will be supplemented with a patient questionnaire specifically designed for breast surgery patients.

All patients will receive the standard preoperative work up, intraoperative procedures, and postoperative care indicated for patients undergoing implant breast reconstruction after mastectomy. Some of these patients will require use of the Alloderm to reconstruct the lower half of the breast pocket. This is already being done by plastic surgeons here at Henry Ford Hospital. The difference will be that the Alloderm tissue matrix used to reconstruct the lower part of the breast pocket for the study patients will have 4 millimeter metallic clips placed in it. Postoperatively these clips will be tracked by ultrasound done in the clinic. As the breast implant is normally expanded by adding saline, we believe the Alloderm matrix will stretch. The movement of these imperceptible clips will be tracked and measured to map the expansion of the matrix in response to the underlying implant stretching the overlying breast pocket and the skin envelope. The pattern of expansion will allow us to develop a mathematical model to describe the stretch pattern of Alloderm matrix used in breast reconstruction. This information will be supplemented with a validated questionnaire specifically designed by breast surgery patients. This will give us both an objective dimensional change in the breast reconstruction as well as a patient-centered evaluation of the reconstruction process.

DETAILED DESCRIPTION:
1. Describe the experimental design/methodology.Prospective consecutive case series.
2. Outline the protocol, corresponding it to the specific aims; identify the data or endpoints to be analyzed to reach the specific aims.

   1. The first 3 candidates will serve as the prototypes for the model. There may be some unanticipated modifications to the setup, patient care, imaging or data analysis. We plan to follow these 3 cases more deliberately and not proceed until all 3 are followed for at least 3 months. After these 3 cases, we anticipate the rest will proceed more smoothly. Placement of the clips to provide the most data is the primary question for these 3 cases.

      The above schematic shows the presumed change is Alloderm size and shape post expansion and corresponding change in location of the vessel clips. The inferior borders is the fixed point. By positioning the clips at regular intervals along the top border, we can measure transverse and horizontal changes. The timing of ultrasound studies is designed to coincide with when these changes are most likely to be visualized during the postoperative period. We may change the dates of the studies. We do not anticipate the the total number of studies will increase because changes after full expansion (completed by postoperative week 4) are slower and smaller in magnitude.
   2. 30 patients enrolled in the study will be studied for position of the metallic markers on postoperative day 1, week 4, month 6, month 12. The location of each clip relative to the fixed anchor point will be recorded and each timepoint. The fixed anchor point is the medial-inner attachment point of the Alloderm® to the chest wall fascia. This is the most inferior/medial point of the Alloderm® tissue matrix. With expansion of the breast expander the chest wall fascia does not move. Only the overlying skin, pectoralis muscle and Alloderm stretch in response to breast prosthesis expansion. We can therefore track movement of the clips embedded in the matrix over time. For each clip we can develop a best fit curve for the 30 subjects studied. This will allow us to develop a mathematical model of the final position and shape of the reconstructed breast at one year out. This model will be compared to existing mathematical models for breast tissue expanders (Mentor Corp.
   3. A standardized validated questionnaire Breast-Q is a patient reported outcomes data instrument. The Breast-Q is conceptually grounded in patient perceptions, able to span the continuum of impact of surgery or validated against appropriate psychometric benchmarks. It allows for quantification of patient satisfaction and health-related quality of life experienced by women undergoing breast surgery. The questionnaire will be administered preoperative, one month postoperative and one year postoperative.

   The BREAST-Q scoring software, QScore, gives clinicians and researchers a simple and accurate way to analyze their data. It features a powerful scoring engine based on RUMM 2020; a data analyzing program developed by Rasch Unidimensional Measurement Models Laboratory in Perth, Australia.

   Each pre and postoperative BREAST-Q module comes with a Microsoft Excel template. The templates help to organize your data for import into the QScore program. Once imported, QScore automatically transforms your raw data into summary scores ranging from 0 (very dissatisfied) to 100 (very satisfied) for each scale.
3. Discuss potential limitations and difficulties in the protocol. Potential limitations include displacement of the vessel clips. If this happens, the patient's results and aesthetic outcome are not compromised. The clips do not cause any harm. These patients will be followed by standard of care protocol but removed from the study.
4. Provide a tentative schedule for conducting and completing this project and, if applicable, the multicenter study.

   The patients will be seen in the office at study enrollment and post surgery at one week, one month, six months and one years for evaluation ultrasound study. The Breast Q questionnaire will be completed preoperatively and then after surgery at one month and one year. one month and one year post surgery. We anticipated all patients enrolled within 6 months of study initiation. Total project should less than 2 years after last patient enrolled.
5. Data collection: Submit a copy of the data collection tool or list the data fields to be collected (review IRB policy, Access to Medical Records for Research on intranet at http://henry.hfhs.org).

Data entry points that will be collected include: The patient's name, age, history of steroid use, past medical history, date of surgery, size of graft used, thickness of the graft used. Also implant size, pre-surgery bra size, distance from each clip to inferiolateral anchor point on ultrasound.

7. DATA ANALYSIS: Describe the analysis of the data and relate this to the specific aims. Describe the statistical analysis in detail (referral to analysis by a multicenter sponsor is not acceptable). The Committee recommends free consultation with the Division of Biostatistics and Research Epidemiology.

There are two types of outcome measurements: the alloderm increased size and stardardized validated questionnaire. We will compare the difference between baseline and each time point after implant. For the alloderm increased size, the student paired-t statistic wil be used to test if there is any stretch in size. For questionnaire outcome, one-sample wilcoxon rank sum test will be used to test the difference in patient satisfication. Bonferrnoi correction is used for multiple comparison and the familywise type I error rate is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

Inclusion of all females from ages 18 and older who undergoing prosthetic breast reconstruction and will require alloderm for lower pole reconstruction.-

Exclusion Criteria:

Exclusion criteria include perioperative radiation. History of allergic reaction to the allograft or its components or the metallic clips.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Develop a mathematical model of the in situ stretch parameters of Alloderm® tissue matrix when used in breast reconstruction. | 18 months

SECONDARY OUTCOMES:
Define patient outcome and expectations with respect to prosthetic breast reconstruction with the use of Alloderm® tissue matrix. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: aamir siddiqui, md, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States